CLINICAL TRIAL: NCT05624567
Title: Symptoms and Quality of Life of Patients With Suspected Endometriosis - a Prospective Multi-center Observational Study
Brief Title: Symptoms and Quality of Life of Patients With Suspected Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, René Wenzl, Ao. Univ. Prof. Dr., Medical University of Vienna
Other Study IDs: 1629/2022
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Endometriosis; Surgery; Pain; Dysmenorrhea; Dyspareunia
MeSH Terms: conditions — Endometriosis; Pain; Dysmenorrhea; Dyspareunia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All patients undergoing surgery due to suspected endometriosis in a previously selected 3-month period within the study period (between 12/2022 and 12/24) (each participating center will define the particular 3 months in question) will be asked to participate in this study. Upon inclusion, patients will be asked to fill out questionnaires regarding endometriosis-associated symptoms as well as a detailed patient history. Furthermore, patients will be asked to fill out 2 standardized questionnaires, one regarding quality of life (Endometriosis-Health Profile-30) and one regarding sexual function (Female Sexual Function Index). Six and 12 months after surgery, patients will again be asked to fill out these two standardized questionnaires as well as a questionnaire regarding postsurgical therapy and endometriosis-associated symptoms. The surgeon will be asked to fill out a form regarding the surgical procedure and possible surgical complications.

The primary endpoints of this multicenter observational study are to prospectively examine:

1. if the individual symptoms correlate with the individual compartments of the surgical #ENZIAN Endometriosis classification
2. if the surgical intervention has an effect on the quality of life in relation to the individual #ENZIAN compartments.

ELIGIBILITY:
Inclusion Criteria:

* Planned surgery for suspected endometriosis
* Age between 18 and 50
* signed informed consent

Exclusion Criteria:

* menopause
* current malignant disease

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Women between 18 and 50 years of age undergoing surgery for suspected endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Symptom correlation with #ENZIAN | 12/2022-12/2024
  Do the individual symptoms correlate with the individual compartments of the surgical #ENZIAN Endometriosis classification
Endometriosis surgery and #ENZIAN - Correlation with quality of life? | 12/2022-12/2024
  Does the surgical intervention have an effect on the quality of life in relation to the individual #ENZIAN compartments.

REFERENCES:
- [Derived] Reiser E, Gobel G, Perricos-Hess A, Buchweitz O, Jaekel M, Westphal E, Rimbach S, Woelfler M, Kraemer B, Kolben T, Pempelfort SD, Pashkunova D, Metzler J, Derihaci RP, Klein P, Janschek E, Guttenberg P, Wuester M, Wolfrum A, Seifert-Klauss V, Enzelsberger SH, Keckstein J, Wenzl R, Seeber B. Evaluation of the association between self-reported pre-operative symptoms with surgically diagnosed endometriosis using the #ENZIAN classification in a multi-centre cohort. Hum Reprod. 2025 Sep 1;40(9):1643-1650. doi: 10.1093/humrep/deaf120. PMID 40682308